CLINICAL TRIAL: NCT02170558
Title: Evaluating Enhanced Metal Reduction Techniques for Definitive CT Scanning to Assess Spinal Fusion With Trabecular Metal Implants (TM-Ardis)
Brief Title: Enhanced Metal Reduction Techniques for Definitive CT Scanning to Assess Spinal Fusion With TM-Ardis
Status: Withdrawn | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSU2013-05S
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Degenerative Disc Disease
Keywords: Trabecular Metal; Metal reduction CT; TM- Ardis
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients implanted w/TM-Ardis: Patients who are receiving a TM-Ardis implant for degenerative disc disease will have a CT scan immediate post op (2 weeks) and again at 6 months to determine if fusion can be assessed with the study metal reduction software. Will utilize TM- Ardis implant and Metal Reduction CT software
  Interventions: Device: TM- Ardis implant and Metal Reduction CT software

INTERVENTIONS:
Device: TM- Ardis implant and Metal Reduction CT software — TM- Ardis implant and Metal Reduction CT software

SUMMARY:
To determine if the subject metal reduction software helps to better visualize bone interphase and fusion reliability. Assess whether the appropriate procedural modification facilitates clearer images when implanted with a trabecular metal spinal implant

DETAILED DESCRIPTION:
To determine if the subject metal reduction software helps to better visualize bone interphase and fusion reliability, and assess whether the appropriate procedural modification facilitates clearer images when implanted with a trabecular metal spinal implant.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent.
* Male or non-pregnant female scheduled for Trabecular Metal (TM - Ardis) implant, single level lumbar.
* Participant must be at least 18 years of age.

Exclusion Criteria:

* Patient is pregnant Patient is unable to comprehend the requirements of the study.
* Patient is unable to undergo scanning (due to body habitus, inability to comply with positioning requirements, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are having a spinal fusion procedure with TM-Ardis and meet the requirements below are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
CT scan to determine if the study software can reduce metal scatter on the scan. | 6 month post operative
  Each CT scan will be evaluated to asses if you can visualize fusion, bone interface, and/or device migration with an experimental metal reduction software for CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Joel Batts, Study Director — Zimmer Biomet Spine
Locations (1):
- St Alphonsus Regional Medical Center, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: Undecided